CLINICAL TRIAL: NCT05045638
Title: A Phase I, Open-label, Fixed Sequence Crossover Study to Investigate the Effect of Coadministration of Sotorasib on the Pharmacokinetics of Rosuvastatin, a Breast Cancer Resistance Protein Substrate, in Healthy Subjects
Brief Title: Effect of Coadministration of Sotorasib on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20200426
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: AMG 510; Sotorasib; Rosuvastatin; Healthy participants
MeSH Terms: interventions — Rosuvastatin Calcium; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin alone (Experimental)
  Interventions: Drug: Rosuvastatin
- Rosuvastatin + sotorasib (Experimental)
  Interventions: Drug: Rosuvastatin; Drug: Sotorasib

INTERVENTIONS:
Drug: Rosuvastatin — Oral dose
Drug: Sotorasib — Oral dose
  Other Names: AMG 510
  Arms: Rosuvastatin + sotorasib

SUMMARY:
A study to determine the effect of sotorasib on the pharmacokinetics (PK) of rosuvastatin, and to assess the PK of rosuvastatin when administered alone, in healthy participants.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects or female subjects, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 30 kg/m2 (inclusive), at the time of Screening.
* Females of nonchildbearing potential

Exclusion criteria:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease, including history of myolysis, not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit - Daytona Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were enrolled at a single center in the United States between 20 August 2021 and 10 October 2021.
Pre-assignment Details: The participants received 10 mg rosuvastatin on Day 1 and 960 mg sotorasib coadministered with 10 mg rosuvastatin on Day 6.
Groups:
- All Participants: On Day 1, rosuvastatin was administered as a single 10 mg dose. On Day 6, sotorasib was administered as a single 960 mg dose and was followed immediately by a single dose of 10 mg rosuvastatin. All participants fasted overnight (at least 10 hours) until 4 hours postdose and refrained from consuming water for 1 hour prior to dosing and 2 hours postdose.
Period: Overall Study
Arm/Group | All Participants
Started | 13
Received Rosuvastatin Alone | 13
Received Rosuvastatin Coadministered With Sotorasib | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of sotorasib or rosuvastatin and had at least 1 postdose safety assessment.
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rosuvastatin
Description: The pharmacokinetic (PK) parameters were determined using standard non-compartmental methods.
Time Frame: Predose (Hour 0), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 hours postdose following administration of rosuvastatin on Days 1 and 6
Population: The PK population included all participants who received at least 1 dose of rosuvastatin or sotorasib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Rosuvastatin: On Day 1, rosuvastatin was administered as a single 10 mg dose. All participants fasted overnight (at least 10 hours) until 4 hours postdose and refrained from consuming water for 1 hour prior to dosing and 2 hours postdose.
- Sotorasib + Rosuvastatin: On Day 6, sotorasib was administered as a single 960 mg dose and was followed immediately by a single dose of 10 mg rosuvastatin. All participants fasted overnight (at least 10 hours) until 4 hours postdose and refrained from consuming water for 1 hour prior to dosing and 2 hours postdose.
Arm/Group | Rosuvastatin | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13 | 13
ng/mL | 3.80 (57.80) | 6.47 (136.00)
Statistical Analysis 1: Comparison: Rosuvastatin vs Sotorasib + Rosuvastatin; The ratios of geometric least squares means (GLSMs) and confidence intervals (CIs) were obtained by taking the exponential of the corresponding differences and CIs on the natural-log (ln) scale; Test type: Other; Ratio of GLSMs = 1.6999, 90% CI 2-sided [1.1860 to 2.4363]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Rosuvastatin
Description: The PK parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Rosuvastatin | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13 | 13
h*ng/mL | 33.20 (57.00) | 44.50 (73.60)
Statistical Analysis 1: Comparison: Rosuvastatin vs Sotorasib + Rosuvastatin; The ratios of GLSMs and CIs were obtained by taking the exponential of the corresponding differences and CIs on the ln scale; Test type: Other; Ratio of GLSMs = 1.3389, 90% CI 2-sided [1.0334 to 1.7347]

3. Primary Outcome: AUC From Time Zero to Infinity (AUCinf) of Rosuvastatin
Description: The PK parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Rosuvastatin | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 12 | 11
h*ng/mL | 36.20 (60.10) | 48.40 (78.90)
Statistical Analysis 1: Comparison: Rosuvastatin vs Sotorasib + Rosuvastatin; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of GLSMs = 1.3382, 90% CI 2-sided [0.9856 to 1.8169]

4. Secondary Outcome: Number of Participants Reporting Any Treatment-Emergent Adverse Events (TEAEs)
Description: Any clinically significant changes in clinical laboratory tests, 12-lead electrocardiograms (ECGs), and vital signs results were recorded as AEs.
Time Frame: Day 1 to Day 41
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

5. Secondary Outcome: Cmax of Sotorasib
Description: The PK parameters were determined using standard non-compartmental methods.
Time Frame: Predose (Hour 0), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on Day 6
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13
ng/mL | 4650 (86.2)

6. Secondary Outcome: AUClast of Sotorasib
Description: The PK parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13
h*ng/mL | 22500 (74.3)

7. Secondary Outcome: AUCinf of Sotorasib
Description: The PK parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sotorasib + Rosuvastatin
Number analyzed (Participants) | 13
h*ng/mL | 22900 (71.7)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 41
Description: The safety population included all participants who received at least 1 dose of sotorasib or rosuvastatin and had at least 1 postdose safety assessment.
Arm/Group | Rosuvastatin | Sotorasib + Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT05045638/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT05045638/SAP_001.pdf